CLINICAL TRIAL: NCT07164976
Title: Phase Ib/II Trial of Ribociclib Plus Anastrozole in Patients With Hormone Receptor-Positive, HER2-Negative Metastatic or Recurrent Breast Cancer
Brief Title: Ribociclib for HR-positive HER2-negative Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nagoya City University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Kazuki Nozawa, Principal Investigator, Nagoya City University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCU-002-Ribo(M)
Record Dates: First submitted 2025-08-23; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; ribociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- phase 1b cohort 1 (Experimental): phase 1b cohort 1
  Interventions: Drug: Ribociclib 400mg
- phase 1b cohort 2 (Experimental): phase 1b cohort 2
  Interventions: Drug: Ribociclib 600mg
- phase 2 part (Experimental)
  Interventions: Drug: Ribociclib 600mg

INTERVENTIONS:
Drug: Ribociclib 400mg — phase 1b cohort 1
  Arms: phase 1b cohort 1
Drug: Ribociclib 600mg — Phase 1b cohort 2
  Arms: phase 1b cohort 2
Drug: Ribociclib 600mg — phase 2
  Arms: phase 2 part

SUMMARY:
This document outlines an investigator-initiated Phase Ib/II clinical trial in Japan, focusing on the combination therapy of ribociclib and anastrozole for patients with hormone receptor-positive (HR-positive), HER2-negative metastatic or recurrent breast cancer. The trial aims to evaluate the efficacy (specifically, overall response rate) and safety of this combination in the Japanese patient population. Nagoya City University is the sponsor of this trial, with funding provided by Novartis Pharma K.K..

Study Design and Endpoints: The trial is structured into two parts:

* Phase Ib: The primary endpoint for this phase is tolerability, which is assessed by dose-limiting toxicities (DLT). Secondary endpoints include pharmacokinetics (PK) of the drugs, as well as the incidence of adverse events (AE) and serious adverse events (SAE).
* Phase II: The primary endpoint for Phase II is the Overall Response Rate (ORR), which will be determined by a blinded central imaging review based on RECIST version 1.1 criteria. Secondary endpoints encompass PK (for the initial 20 patients), ORR as assessed by the investigator, progression-free survival (PFS), overall survival (OS), and the overall incidence of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer.
* Hormone receptor-positive (ER positive and/or PgR positive) and HER2-negative disease:

ER positive: ≥1% positive cells or Allred score ≥3.

PgR positive: ≥1% positive cells or Allred score ≥3.

HER2 negative: IHC 0, 1+, or 2+ with no ISH amplification.

* Advanced or recurrent breast cancer (unresectable, recurrent, or Stage IV).
* Age ≥18 years at registration.
* ECOG Performance Status of 0-1.

Exclusion Criteria:

* Symptomatic visceral metastases or deemed unsuitable for endocrine therapy.
* Prior endocrine therapy or chemotherapy for metastatic/recurrent disease.
* Prior CDK4/6 inhibitor exposure (perioperative or metastatic setting).
* Adjuvant endocrine therapy within 35 days before study start.
* Active malignancy other than allowed exceptions (e.g., resected skin cancers, ≥5-year disease-free cancers).
* Hypersensitivity to ribociclib, anastrozole, or their components (including soy/peanut allergy, sugar intolerances).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1b part: Dose Limiting Toxicity | From enrollment to the end of treatment at 4 weeks
Phase 2 part: Overall response rate | From enrollment to the end of treatment at 24 weeks

SECONDARY OUTCOMES:
Phase 1b part: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From enrollment to the end of treatment at 4 weeks
Phase 1b part: Peak Plasma Concentration (Cmax) | From enrollment to the end of treatment at 4 weeks
Phase 2 part: Overall Response Rate | From enrollment to the end of treatment at 24 weeks
Phase 2 part: PFS | Time Frame: From enrollment to the end of treatment at 24 weeks
Phase 2 part: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From enrollment to the end of treatment at 24 weeks

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol